CLINICAL TRIAL: NCT00310739
Title: Urinary Marker for Oxidative Stress in Human Cisplatin- Induced Renal Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Other Study IDs: 16-50
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-04

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
We previously reported early measurement of urinary MDA might be a useful marker for the prediction of CDDP-induced renal damage in rat. The purpose of this clinical study is to test whether the changes of human urinary excretion of MDA, and can be used as early biomarker for the prediction of development of CDDP-induced ARF.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients have neck cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Tsuji, MD, Principal Investigator — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan